CLINICAL TRIAL: NCT05928442
Title: Interest of Salivary Signature of Endometriosis in the Heathcare Pathway of Adolescent - The ADOmiARN Study
Brief Title: Interest of Salivary Signature of Endometriosis in the Heathcare Pathway of Adolescent
Acronym: ADOmiARN
Status: Recruiting | Type: Observational
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry); iGenSeq (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-02
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis
Keywords: miRNA; RNA; Machine learning algorithms; Adolescents
MeSH Terms: conditions — Endometriosis | interventions — Reagent Kits, Diagnostic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- "Endometriosis" patients: Patient with a formal endometriosis diagnosed by clinical examination and imaging.
  At least 20 patients
  Interventions: Device: in vitro diagnostic medical device; Behavioral: Completion of a self-questionnaire
- "Discordants" patients: Patient with suspected endometriosis for whom the diagnosis is the source of a discrepancy between clinical examination and imaging data, AND a surgical indication.
  At least 20 patients
  Interventions: Device: in vitro diagnostic medical device; Behavioral: Completion of a self-questionnaire
- "Surgery" patients: Patient with a gynaecological indication for surgery of the small pelvis AND symptoms suggestive of endometriosis.
  At least 20 patients
  Interventions: Device: in vitro diagnostic medical device; Behavioral: Completion of a self-questionnaire

INTERVENTIONS:
Device: in vitro diagnostic medical device — Collection of 2 saliva samples at inclusion.
Behavioral: Completion of a self-questionnaire — Completion of a self-questionnaire on symptom and quality-of-life at inclusion.
Device: in vitro diagnostic medical device — Collection of 1 saliva sample at the follow-up visit.
  Groups: "Discordants" patients; "Surgery" patients

SUMMARY:
ADOmiARN is a multicentre, prospective, longitudinal, non-interventional, observational study carried out in obstetrics, gynecology and pediatrics departments in France and in Belgium.

The main objective is to confirm the interest of the in vitro diagnostic medical device (EndoTest®) in adolescents with suspected endometriosis.

The study population is made up of females aged 10 to 19 years with formally diagnosed endometriosis or suspected endometriosis.

The patients concerned by the study are managed without any change in the care pathway, no any change in the therapeutic indications, no any change in the diagnostic examinations (imaging or biology) required according to the context, which are carried out in accordance with the national guidelines.

In this study, the management and follow-up of patients :

* Are not imposed by the study: the doctor remains free to make medical prescriptions (treatments and examinations) and to determine the interval between consultation visits,
* Are not modified in comparison with the usual follow-up, except for the performance of :

  * Collection of saliva
  * Completion of a self-questionnaire on symptom and quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 10 and 19 years,
* Patient over 18 or legal representatives of patient under 18 who has dated and signed the consent form,
* Patient with pelvic MRI available and conduct within 12 months prior to inclusion,
* Patient from one of the 3 study populations:

  * A formal endometriosis diagnosed by clinical examination and imaging or
  * With prescription for coelioscopy because of a discrepancy between clinical and radiological findings or
  * A surgical indication for a pathology of the small pelvis other than endometriosis, in adolescents with suspected endometriosis faced with symptoms suggestive (dysmenorrhea, chronic or cyclic pelvic pain, urinary disorders cycle-dependent)
* Patient affiliated to the healthcare system.

Exclusion Criteria:

* Known pregnancy in progress,
* Known infection with the human immunodeficiency virus (HIV),
* Personal history of cancer,
* Adolescent subject to a protective measure or placed adolescent,
* Adolescent or her legal representatives presenting important difficulties in reading French language,
* Patient or her legal representatives who have objected to the collection of her data,
* Patient participating in an interventional study with drug or medical device or in the exclusion period of an interventional study
* Patient who has participated or is participating in another study evaluating miRNA in endometriosis.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population made up of 3 differents adolescents populations:
  * "Endometriosis" patients: diagnosis confirmed by imaging; endometriosis formally diagnosed on clinical or imaging examination (ovarian endometriosis and/or severe deep endometriosis with vaginal, lateral or colorectal involvement)
  * "Discordants" patients: surgical confirmation; suspected endometriosis with discordant clinical and radiological data requiring surgical care (exploratory coelioscopy) for diagnosis in routine care, based on national recommendations and after validation by in RCP
  * "Sugery" patients: Surgical procedure motivated by a reason other than endometriosis: adolescents with another pelvic pathology requiring a planned surgical procedure, whether or not related to suspected endometriosis (ovarian cyst, uterine malformation) and with evocative symptoms of endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of adolescents with a negative EndoTest® despite a validated diagnosis of endometriosis by coelioscopy or other surgical movement (false negative). | Through the end of study inclusions, an average of 1 year
  Confirm the interest of EndoTest® in adolescents with suspected endometriosis

CONTACTS AND LOCATIONS:
Locations (13):
- Hôpital de la Citadelle, Liège, Belgium
- France (11):
  - Centre chirurgical L'Avancée, Aix-en-Provence
  - CHU Angers, Angers
  - Clinique Tivoli-Ducos, Bordeaux
  - CHU Caen, Caen
  - AP-HM Hôpital de la Conception, Marseille
  - CHU Caremeau, Nîmes
  - Hôpital Tenon, Paris
  - APHP, Hôpital Cochin Port Royal, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
- Universitätsklinik für Frauenheilkunde, Inselspital Bern, Bern, Switzerland